CLINICAL TRIAL: NCT00230048
Title: Interactive Motivational Media for Perinatal Drug Abuse
Brief Title: Interactive Motivational Media for Perinatal Drug Abuse - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-14621-3; R21DA014621 (NIH)
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assessment only (No Intervention)
- Brief intervention (Experimental)
  Interventions: Behavioral: Brief computer-delivered intervention

INTERVENTIONS:
Behavioral: Brief computer-delivered intervention — Brief (20-minute) computer delivered intervention, plus two subsequent non-tailored mailings.
  Arms: Brief intervention

SUMMARY:
Interactive Motivational Media for Perinatal Drug Abuse

DETAILED DESCRIPTION:
The goal of this exploratory/developmental proposal is to develop a low-cost, highly adaptable brief motivational intervention for perinatal drug abuse via embedding motivational principles in a self-contained interactive computer system. The Motivation Enhancement System (MES) will utilize a touch-screen, audio enhancement, and an interactive narrator to guide women in the immediate post-partum period through evaluation (thus facilitating self-report) and a one-time motivational intervention. A taxi voucher will be provided to further facilitate entry into treatment, and multiple tailored self-help mailings will be issued following discharge. If validated, this intervention could offer a highly cost-effective, replicable, and prescriptive method for increasing self-change and treatment involvement in drug abusers. Following development of the MES, a preliminary pilot phase will study the use of the MES with post-partum drug-using women and make necessary modifications, using data from participant debriefings and a single-case research design. After optimization of the MES, a clinical trial will randomly assign 120 post-partum drug-using women into treatment or assessment only conditions, with a 3-month blinded follow up to evaluate intervention effects on drug use and treatment involvement. Toxicological and self-report measures, as well as objective analysis of infant development, will be utilized. Participants will be lower socioeconomic status urban women.

ELIGIBILITY:
Woman in immediate postpartum period

Inclusion Criteria:

Screen positive for drug use (self-report)

Exclusion Criteria:

Frank psychosis or other cognitive impairment, fatigue, grief over medically compromised infant, inability to communicate in English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2001-09; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Ondersma, Ph.D., Principal Investigator — ACT
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Result] Ondersma SJ, Chase SK, Svikis DS, Schuster CR. Computer-based brief motivational intervention for perinatal drug use. J Subst Abuse Treat. 2005 Jun;28(4):305-12. doi: 10.1016/j.jsat.2005.02.004. PMID 15925264
- [Result] Ondersma SJ, Svikis DS, Schuster CR. Computer-based brief intervention a randomized trial with postpartum women. Am J Prev Med. 2007 Mar;32(3):231-8. doi: 10.1016/j.amepre.2006.11.003. Epub 2007 Jan 22. PMID 17236741

RESULTS

PARTICIPANT FLOW:
Groups:
- Assessment Only: This arm answered questions only, but received no intervention.
- Brief Intervention: Brief computer-delivered intervention following motivational approach, adapted from Motivational Interviewing: Decisional balance, normed feedback, and optional goal-setting.
Period: Overall Study
Arm/Group | Assessment Only | Brief Intervention
Started | 52 | 55
Completed Intervention/Control Session | 52 | 55
Completed | 39 | 37
Not Completed | 13 | 18
Not completed — Lost to Follow-up | 13 | 18

BASELINE CHARACTERISTICS:
Groups:
- Brief Intervention: Brief computer-delivered intervention following 5As/5Rs approach.
- Total: Total of all reporting groups
Arm/Group | Assessment Only | Brief Intervention | Total
Number analyzed (Participants) | 52 | 55 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 55 | 107
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.2 (5.4) | 25.9 (5.7) | 25.1 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 107
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 55 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug Use at 3 Months
Description: The number of participants postive for drug use using participant's self-report of drug use and urinalysis. Participants were considered positive if self-report and/or urinalysis were positive.
Time Frame: 3 months
Population: Intent to treat, treating participants lost to follow-up as positive.
Measure: Number; unit: participants
Groups:
- Assessment Only: Assessment only, via computer.
- Brief Intervention: Assessment plus 20-minute interactive session with computer, designed to be maximally similar to a therapist-delivered motivational session.
Arm/Group | Assessment Only | Brief Intervention
Number analyzed (Participants) | 52 | 55
participants | 49 | 48

2. Primary Outcome: Treatment Engagement
Description: Completing at least a single intake or treatment session of any kind, focused on substance use within the previous 3 months.
Time Frame: 3 months
Population: ITT, treating all participants lost to follow up as failures (i.e., not receiving any treatment services)
Measure: Number; unit: participants
Arm/Group | Assessment Only | Brief Intervention
Number analyzed (Participants) | 52 | 55
participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Assessment Only | Brief Intervention
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/55
Other Adverse Events (participants affected / at risk) | 0/52 | 0/55

LIMITATIONS AND CAVEATS:
Generalizability limited by relatively small sample, attrition of 29%, and restriction to low-income mothers. Second, power limitations prevented verification of effects on the dichotomous outcomes, despite effects in the small-moderate range.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No